CLINICAL TRIAL: NCT01106118
Title: Therapeutic Effectiveness of Vardenafil in ED Patients With the Metabolic Syndrome in Daily Clinical Practice
Brief Title: Therapeutic Effectiveness of Vardenafil in Patients With Erectile Dysfunction and Metabolic Syndrome in Daily Clinical Practice
Acronym: REVITALISE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14872; LV0901 (Other: Company internal)
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Vardenafil (Levitra, BAY38-9456)

INTERVENTIONS:
Drug: Vardenafil (Levitra, BAY38-9456) — Patients with diagnosis of erectile dysfunction and metabolic syndrome who get vardenafil in routine treatment as prescribed by physician

SUMMARY:
The primary goal of this international non-interventional study is to investigate the therapeutic effectiveness of vardenafil (film-coated tablet) in Erectile Dysfunction patients with the Metabolic Syndrome in daily clinical practice. It will include a large number of patients with various underlying conditions with different cultural and demographic backgrounds from different geographic areas.

ELIGIBILITY:
Inclusion Criteria:

* Erectile Dysfunction (ED) patient who has newly been prescribed vardenafil (Levitra film-coated tablet) in accordance with the terms of the local marketing authorization.
* Diagnosis of erectile dysfunction at the discretion of the physician, based on the patients ED history.
* No use of any Phosphodiesterase Type 5 (PDE5) inhibitor within 1 month of study entry.
* Documented Metabolic Syndrome (MetS), preferably according to the definition of the International Diabetes Foundation.

Exclusion Criteria:

* Do not follow the contraindications and warnings of the Summary of Product Characteristics.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of erectile dysfunction and metabolic syndrome who get vardenafil in routine treatment
Sampling Method: Non-Probability Sample
Enrollment: 2289 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with a clinically relevant, intra-individual improvement in erectile function defined as an increase of 4 points in the erectile function domain of the International Index of Erectile Function (IIEF) | After approx 12 weeks

SECONDARY OUTCOMES:
Patients with an increase of 5 points in the Erectile Dysfunction domain of the IIEF after approx. 12 weeks | After approx. 12 weeks
Subjects with normal erectile function (IIEF-EF ³26) After approx. 12 weeks | After approx. 12 weeks
Subjects with mild Erectile Dysfunction (IIEF-EF 22-25) After approx. 12 weeks | After approx. 12 weeks
Optional by country, the effect of vardenafil on health-related quality of life (HRQoL) using the Aging Males Symptoms (AMS) Scale | After approx. 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- Many Locations, Egypt
- Many Locations, Israel
- Many Locations, Kazakhstan
- Many Locations, Kyrgyzstan
- Many Locations, Lebanon
- Many Locations, Russia
- Many Locations, Saudi Arabia
- Many Locations, Singapore
- Many Locations, South Korea
- Many Locations, Ukraine

REFERENCES:
- [Result] Shabsigh R, Mattern A; REVITALISE Study Group. REVITALISE: A Large Observational Study Assessing the Safety and Effectiveness of Vardenafil in Men With Erectile Dysfunction and Metabolic Syndrome. Sex Med. 2016 Sep;4(3):e135-44. doi: 10.1016/j.esxm.2016.03.027. Epub 2016 Apr 14. PMID 27151768